CLINICAL TRIAL: NCT06774287
Title: Evaluation of the Karman Line Memory Strategy Training, a Combined Computerized and Face-to-face Compensatory Treatment Targeting Memory Complaints After Acquired Brain Injury, Using Single-case Experimental Design Methodology
Brief Title: Evaluation of the Karman Line Memory Strategy Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Klimmendaal Revalidatiespecialisten (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KNP23PROJ1
Record Dates: First submitted 2024-09-25; First posted 2025-01-14 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Acquired Brain Injury (Including Stroke)
Keywords: Compensatory brain games; Acquired Brain Injury; memory disorder
MeSH Terms: conditions — Brain Injuries; Memory Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment as usual (Active Comparator): Treatment as usual contains 10 memory strategy sessions (two sessions per week) with a therapist in the rehabilitation centre.
  Interventions: Behavioral: Treatment as usual
- Karman Line memory training (Experimental): Karman Line memory strategy training contains 6 weekly memory strategy sessions in the rehabilitation centre, combined with practicing digital games at home and using a memory app.
  Interventions: Behavioral: Karman Line memory strategy training

INTERVENTIONS:
Behavioral: Karman Line memory strategy training — The memory strategy training consists of six weekly face-to-face treatment sessions. After sessions 3-5, the participant will play 8 levels in total of the Karman Line memory game on their computer or mobile device. In these levels they practice the strategies that are introduced in the face-to-face treatment in a safe digital environment. Also, the Karman Line memory app is provided.
  Arms: Karman Line memory training
Behavioral: Treatment as usual — Treatment as usual contains ten sessions, with nine obligatory sessions supplemented with 1 (of five) non-obligatory sessions. Which non-obligatory sessions is chosen is dependent on the patients treatment goals.
  Arms: treatment as usual

SUMMARY:
Rationale: Acquired brain injury (ABI) often results in memory deficits that can have a big impact on social and vocational functioning of patients. Rehabilitation treatment of memory dysfunction consists of optimizing memory performance by using effective compensation strategies. Several effective memory-strategy training programs have been developed. However, these often contain labor-intensive treatment protocols that are possibly an overtreatment of ABI patients with relatively mild memory impairments. On the other hand there is a sprawl of commercial computerized cognitive training programs or 'brain games' available that claim to restore memory function. However, research has repeatedly shown that treatment effects of available brain games do not generalize to daily life functioning. With the shortcomings of current memory treatment programs in mind, the investigators developed a combined computerized and face-to-face training of memory strategies, which consists of a shortened traditional face-to-face treatment combined with an innovative Brain Game based on compensation strategies instead of restorative training. This is a promising cost-effective intervention that provides the possibility of repeated practice at home to train compensatory strategies in a safe and imaginative digital environment. The hypothesis is the strategy training will promote generalization, also after rehabilitation ends.

Objective: The primary objective is the evaluation of the potential positive effect of the combined computerized and face-to-face memory treatment on effective memory strategy use and reducing subjective memory failures in ABI patients with memory deficits in the chronic phase of acquired brain injury (>3 months after injury).

Study design: The study will be a multiple-baseline across individuals single-case experimental design (SCED). Three patients will receive treatment as usual and three patients will receive a shortened treatment combined with the game, which will be referred to as the 'Karman Line memory strategy training'.

Study population: The study population consists of patients referred for outpatient cognitive rehabilitation. Participants eligible for the study must have memory deficits and complaints due to Acquired Brain Injury (ABI) of nonprogressive nature (i.e. TBI, stroke), with a minimum time post-onset of 3 months. Age has to be between 18 and 75 and participants have to live independently at home. Memory deficits will be assessed by neuropsychological examination, memory complaints will be assessed by the Everyday Memory Questionnaire-Revised (EMQ-R). In one year six to eight participants will be recruited.

Intervention: The Karman Line memory strategy training consists of six weekly treatment sessions under the guidance of a therapist. The protocol is a shortened version of an existing memory strategy training (treatment as usual), which contains ten sessions. In the sessions, patients get information about memory and memory strategies and learn to apply those to their personal treatment goals. Inbetween the sessions, the participant will work on personal memory goals and practice the strategies by playing the corresponding levels of the memory game at home.

Main study parameters/endpoints: The main study parameter is the three most commonly reported memory complaints selected from the 13-item scale of the EMQ-R. The primary outcome measure is not the EMQ-R, but a personalized set of measurement VAS-scales for each patient. Secondary study parameters include the impact of memory problems on activities and participation, the achievement of personalized treatment goals, objective strategy use, objective memory functioning, metacognitions about memory and measures of feasibility by patients and practitioners.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The burden in the study consists of participating in repeated measurements, therapy sessions, and homework assignments. All tests and methods that are used are non-invasive and not stressful for the patient. All tests and tasks will be based on widely-used validated and reliable paper-pencil or computer tasks. Treatment is non-invasive and scarcely stressful: a therapist will always be present and assess the patient's burden and eventually take appropriate measures such as inserting a resting break.

ELIGIBILITY:
Inclusion criteria:

* presence of subjective memory complaints. Memory complaints will be operationalized as ≥1 standard deviation on the total score of the EMQ-R questionnaire in comparison with the healthy control norm.
* presence of mild to moderate objective memory deficits, objectified with neuropsychological assessment for clinical purposes. Mild to moderate memory deficits will be operationalized as test score ≥1 standard deviation (SD) and <2 SD in comparison to the normative mean on at least two separate memory measures and no more than one measure ≥ 2SD. For each task the norm data that is described in the test manual will be used.
* Age: 18-75 years
* Non-progressive acquired brain injury
* Minimal time post-onset of 3 months
* Outpatient rehabilitation
* Living independently at home
* Premorbid functioning: score 4 on the Verhage scale

Exclusion criteria:

* Severe memory deficits
* Inability to speak and/or understand the Dutch language
* Severe disorders in executive functioning
* Severe psychiatric problems
* Neurodegenerative disorders
* Substance abuse
* Aphasia
* Neglect
* No access to a smartphone and a tablet/laptop with internet connection
* Unable to look at a computer screen for 15 minutes
* Unable to operate a keyboard or computer mouse.
* No informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
memory complaints | every other day during 8-10 weeks, weekly during 3-5 weeks
  The 13-item scale of the everyday memory questionnaire-revised (EMQ-R) is used to select the three most common memory complaints that are targeted with the intervention. The primary outcome measure is not the EMQ-R, but a personalized set of measurement visual analogue scales (VAS) for each patient. The total score (range 0-30) will be used as outcome measure. A higher score indicates more memory complaints, which is a worse outcome.

SECONDARY OUTCOMES:
The impact of memory problems on activities and participation | every other day during 8-10 weeks, weekly during 3-5 weeks
  visual analogue scale (range 0-10), 10 meaning more impact on activities and participation
The achievement of personalized treatment goals | 4 measurements during study participation (during 13 weeks)
  The achievement of personalized treatment goals is measured by goal attainment scaling (GAS). GAS is a mathematical technique for quantifying the achievement of goals set, used in rehabilitation. GAS is described as a method of scoring the extent to which a patient's individual goals are achieved in the course of intervention. In effect, each patient has their own outcome measure, but this is scored in a standardized way. The achievement of each goal can be measured on a 5-point scale ranging from -2 to +2. Outcomes can be quantified in a single aggregated Goal Attainment Score. This method gives a numerical T-score which is normally distributed about a mean of 50 (if the goals are achieved precisely) with a standard deviation of around this mean of 10 (if the goals are overachieved or underachieved). Goals are individually identified to suit and the levels are individually set around their current and expected levels of performance.
Objective strategy use task | 4 measurements during study participation (during 13 weeks)
  The original strategy observation task (SOT )is developed to observe strategy use during a memory task that mimics daily life situations. For repeated measurements, parrallel versions are used. Participants are instructed to remember a story that was played as an audio clip. Additionally, participants are asked to spontaneously recall the story exactly 5 min after the end of the audio clip. In the meantime, they are instructed to solve basic math problems. The instructions emphasize that participants should remember as much information as possible and that they are allowed to do or use anything to help them remember the information. The strategic behavior of the participants is recorded on an observation list.
  For analyses, the total number of strategies on the SOT is used, including both observed and self-reported strategies.
Rivermead Behavioural Memory Test-3 (RBMT-3-NL) | 2 measurements during study participation (during 13 weeks)
  The RBMT-3-NL is a valid ecologically valid memory batty that is usable for repeated measurement of memory. An overall General Memory Index can also be derived which has a mean of 100 and standard deviation of 15.
Location Learning Test (LLT) | 2 measurements during study participation (during 13 weeks)
  The LLT is a test that can be used to measure episodic spatial memory for object locations. Normalized scores for immediate and delayed spatial memory are computed (percentiles 0-100).
Verbal learning and memory test (VLGT). | 2 measurements during study participation (during 13 weeks)
  The VLGT is the Dutch translation of the internationally widely used Californian Verbal Learning Test (CVLT) and is designed to assess encoding, recall, and recognition of auditory-verbal information. Normalized scores for immediate and delayed verbal memory are computed (percentiles 0-100).
Delis-Kaplan Executive Function System Color Word Interference Test (D-KEFS CWIT) | 2 measurements during study participation (during 13 weeks)
  The D-KEFS CWIT contains measures of attention and information processing speed (conditions 1 and 2) and executive functioning, more specifically inhibition and cognitive flexibility (conditions 3 and 4). Normalized standard scores can be computed (range 0-19, mean: 10, standard deviation: 3).
Wechsler Memory Scale IV-NL Symbol span | 2 measurements during study participation (during 13 weeks)
  Symbol span is a measure of visual working memory. Normalized standard scores can be computed (range 0-19, mean: 10, standard deviation: 3).
Wechsler Adult Intelligence Scale IV-NL digit span (WAIS-IV-NL DS) | 2 measurements during study participation (during 13 weeks)
  The digit span is a measure of verbal working memory. Normalized standard scores can be computed (range 0-19, mean: 10, standard deviation: 3).
Cognitive Failure Questionnaire (CFQ) | 4 measurements during study participation (during 13 weeks)
  The CFQ is a commonly used self-report measure of cognitive errors experienced in daily life . The questionnaire consists of 25 items, rated on a 5-point scale (range 0-125, higher score meaning more cognitive errors). Four additional questions inform on potential increases in the occurrence of these mistakes and the extent to which an individual finds these experiences troublesome, annoying, or worrisome.
Strategy Use in daily life Inventory (SUI) | 4 measurements during study participation (during 13 weeks)
  The SUI measures strategy use in daily life with two subscales. The subscale External Strategies consists of 6 items and includes the use of memory aids, such as taking notes or using a calendar. The subscale Internal Strategies consists of 8 items and includes mnemonics such as mental rehearsal or creating associations. Participants indicate how often they use a certain strategy by rating items on a 5-point Likert scale. Average item scores were calculated for each subscale (external strategies range 0-30, internal strategies range 0-40, higher score meaning more strategies used).
Adapted Illness Cognition Questionnaire (ICL) | 4 measurements during study participation (during 13 weeks)
  The ICL measures illness cognitions that are assumed to be an important mediator between disease and patients' well-being . The two subscales 'helplessness' and 'acceptance' each consist of 6 items. No total score can be computed, average item scores were calculated for each subscale (range 0-24, higher scores reflecting more experienced helplessness (subscale 1) and more acceptance (subscale 2)). The questionnaire will be adapted so that it can be used to measure cognitions regarding 'memory complaints' instead of cognitions regarding illness in general
Measure of feasibility by patients and practitioners 1: qualitative questionnaire | 1 measurement during study participation (during 13 weeks)
  The subjective effectiveness and feasibility of the whole Karman Line memory strategy training intervention will be measured by a qualitative questionnaire that is completed by the therapist and patient after the intervention.
Measure of feasibility by patients and practitioners 2: the System User Scale | 1 measurement during study participation (during 13 weeks)
  The questionnaire consists of 10 items, rated on a 5-point scale (range 0-50, higher score meaning better game user expercience)
Measure of feasibility by patients 3: time spent playing the game | during study participation (during 13 weeks)
  Time spent on playing the different levels of the game and mistakes that are made while playing, which will be monitored automatically.
Measure of feasibility by patients 4: number of dropouts and no shows | during study participation (during 13 weeks)
  * The number of, and reasons for, dropouts during the intervention
  * The number of, and reasons for, no-shows of the face-to-face sessions

CONTACTS AND LOCATIONS:
Locations (1):
- Klimmendaal Revalidatiespecialisten, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided